CLINICAL TRIAL: NCT04339608
Title: A Prospective, Longitudinal, Observational Study of Healthcare Workers and the General Population to Watch for Flu-like Symptoms in Suspicion of COVID 19
Brief Title: Max COVID19- Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Max Healthcare Insititute Limited (Other)
Responsible Party: Sponsor
Other Study IDs: Covid-19/MHC/2020
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In view of the increasing cases of COVID-19 in India and the possibility of the exponential rise of the cases, this study has been designed to collect data of the healthcare workers of Max Hospital and the general population. Our objective is to identify individuals with flu-like symptoms in suspicion of COVID-19 and follow them weekly up to 8 weeks until the pandemic resolves. The data will be collected through an online questionnaire circulated via Emails or WhatsApp.

DETAILED DESCRIPTION:
The primary objective of this study is to screen and identify individuals with flu-like symptoms and follow-them up weekly. In the study, baseline data will be collected online and then weekly follow up will be done with the participants for 4 weeks via opted communication method. There will be no physical contact and we are also avoiding the use of papers so as to avoid possible transmission. Participation in this study will be entirely voluntary and the questionnaire will be accessible to the participants only when they mark "Agree" on the form.

The data collection form is available in English and Hindi.

The study questionnaire includes questions related to general health status, clinical symptoms, Food security, and job security.

ELIGIBILITY:
Inclusion Criteria:

* Indian males and females currently living in India, OR
* All the employees of Max Super Speciality Hospital, New Delhi, India

Exclusion Criteria:

* Anyone who has filled the questionnaire once per household

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include all the healthcare workers of Max Super Speciality Hospital, New Delhi, India, and all males and females from the general population. One questionnaire will be filled up per household.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 positive case | 4-8 weeks
  An individual identified with the clinical symptoms when tested positive for COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Sujeet Jha, MRCP (U.K), Principal Investigator — Max Healthcare
Locations (1):
- Max Super Speciality Hospital, A Unit of Devki Devi Foundation, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing protocol is undecided at this stage. We may, however, provide the data if requested.

REFERENCES:
- [Derived] Jha S, Soni A, Siddiqui S, Batra N, Goel N, Dey S, Budhiraja S, Naithani R. Prevalence of Flu-like Symptoms and COVID-19 in Healthcare Workers from India. J Assoc Physicians India. 2020 Jul;68(7):27-29. PMID 32602677